CLINICAL TRIAL: NCT07388797
Title: Impact of Serum Progesterone Levels on Embryo Transfer Day on Clinical Pregnancy in Frozen-thawed Embryo Transfer Cycles Using Hormone Replacement Therapy: a Prospective Observational Study
Brief Title: Impact of Serum Progesterone Levels on Embryo Transfer Day on Clinical Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2025.875
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Reproductive Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypotheses:

We hypothesize that serum progesterone levels on the day of embryo transfer in HRT-FET cycles are positively associated with clinical pregnancy rates.

Aims:

To evaluate the relationship between serum progesterone levels on embryo transfer day and clinical pregnancy outcomes in frozen-thawed embryo transfer cycles using hormone replacement therapy (HRT).

Primary outcome:

To compare the incidence of clinical pregnancy outcome in those infertility patients undergoing frozen embryo transfer with caterized Progesterone level on the day of embryo transfer

Secondary outcomes:

Biochemical pregnancy rate. Implantation rate. Early pregnancy loss rate. Ectopic pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing FET cycles
* Infertility patients aged >18 years old and < 42 years old
* BMI < 30 kg/m2
* Transfer of at least one good-quality embryo.

Exclusion Criteria:

* Severe endocrine disorders (e.g., thyroid dysfunction, premature ovarian failure).
* Severe uterine factors without treatment (severe endometriosis, extensive or subendometrial fibroid, uterine adherent, endometrial polyps)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All infertility patients undergoing FET at the Assisted Reproductive Technology Unit of the department of Obstetrics and Gynecology in the Prince of Wales Hospital
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate (CPR) | 6 weeks of gestation and ultrasound scanning will be performed to confirm at least one gestational sac around 1 to 3 months after FET
  Rate of clinical pregnancy outcome in subjects undergoing FET

SECONDARY OUTCOMES:
Biochemical pregnancy rate | Up to 12 weeks
  Rate of biochemical pregnancy outcome in subjects undergoing FET
Implantation rate | Up to 12 weeks
  Rate of implantation in subjects undergoing FET
Early pregnancy loss rate | Up to 12 weeks
  Rate of early pregnancy loss in subjects undergoing FET
Ectopic pregnancy rate | Up to 12 weeks
  Rate of Ectopic pregnancy in subjects undergoing FET

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided